CLINICAL TRIAL: NCT05620147
Title: Effect of Apical Third Enlargement to Different Preparation Sizes and Tapers of EdgeFile X7 on Postoperative Pain and Intra-canal Bacterial Reduction in Patients With Necrotic Pulp: A Randomized Clinical Trial
Brief Title: Effect of Apical Enlargement to Different Preparation Sizes and Tapers on Pain and Bacterial Reduction in Necrotic Pulp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen AwadAllah Abbas Ibrahim, Lecturer Assisstant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2/11/2022
Record Dates: First submitted 2022-11-02; First posted 2022-11-17 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Necrotic Pulp
Keywords: Apical enlargement; Postoperative pain; Intra-canal bacterial reduction; Preparation taper; EdgeFile X7
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Root canal instrumentation EdgeFile X7 to size #35/0.06 (Experimental): The mechanical preparation will be continued using EdgeFile X7 #35 .04 and #35 .06
  Interventions: Other: Root canal instrumentation EdgeFile X7 to size #35/0.06
- Root canal instrumentation EdgeFile X7 to size #45/0.04 (Experimental): The mechanical preparation will be continued using EdgeFile X7 #35 .04, #40 .04 and #45 .04
  Interventions: Other: Root canal instrumentation EdgeFile X7 to size #45/0.04
- Root canal instrumentation EdgeFile X7 to size #45/0.06 (Experimental): The mechanical preparation will be continued using EdgeFile X7 #35 .04, #40 .04, #45 .04 and #45 .06
  Interventions: Other: Root canal instrumentation EdgeFile X7 to size #45/0.06
- Root canal instrumentation EdgeFile X7 to size #35/0.04 (Active Comparator): The mechanical preparation will be continued using EdgeFile X7 #35 .04
  Interventions: Other: Root canal instrumentation EdgeFile X7 to size #35/0.04

INTERVENTIONS:
Other: Root canal instrumentation EdgeFile X7 to size #35/0.06 — Instrumentation will be performed using an endodontic motor at a speed of 300 rpm and a torque of 2 Ncm
  Other Names: EdgeEndo
  Arms: Root canal instrumentation EdgeFile X7 to size #35/0.06
Other: Root canal instrumentation EdgeFile X7 to size #45/0.04 — Instrumentation will be performed using an endodontic motor at a speed of 300 rpm and a torque of 2 Ncm
  Other Names: EdgeEndo
  Arms: Root canal instrumentation EdgeFile X7 to size #45/0.04
Other: Root canal instrumentation EdgeFile X7 to size #45/0.06 — Instrumentation will be performed using an endodontic motor at a speed of 300 rpm and a torque of 2 Ncm
  Other Names: EdgeEndo
  Arms: Root canal instrumentation EdgeFile X7 to size #45/0.06
Other: Root canal instrumentation EdgeFile X7 to size #35/0.04 — Instrumentation will be performed using an endodontic motor at a speed of 300 rpm and a torque of 2 Ncm
  Other Names: EdgeEndo
  Arms: Root canal instrumentation EdgeFile X7 to size #35/0.04

SUMMARY:
The aim of this prospective randomized clinical trial is to evaluate the effect of different apical size and taper preparation (35. 04; 35. 06; 45. 04 and 45. 06) on postoperative pain at 6, 12, 24, 48 and 72 hours, and intra-canal bacterial count in patients having mandibular premolars with necrotic pulps.

DETAILED DESCRIPTION:
* Patients will be clinically and radiographically examined and their eligibility will be assessed. Eligible patients will be treated in one visit.
* Patients will be randomly assigned to one of 4 groups: experimental groups of root canal instrumentation with EdgeFile X7 to size #35/0.06 or #45/0.04 or #45/0.06 or the comparator group to size #35/0.04. Intra-canal bacterial count will be measured using a culture technique. Bacterial samples will be taken before and after root canal instrumentation. After endodontic treatment, patients will be given postoperative instructions and informed, in case of pain, to receive ibuprofen 400 mg as rescue medication.
* Postendodontic pain intensity and incidence at the different pain categories (No, mild, moderate, severe) will be assessed at 6, 12, 24, 48 and 72 hours postoperatively using Numerical Rating Scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients, American Society of Anesthesiologists (ASA) I and II.
* Patient's age ranges between 18 to 35 years with no sex predilection.
* Patients with single-rooted mandibular premolars with asymptomatic necrotic pulp.
* Patients who can understand the Numerical Rating Scale (NRS).
* Patients able to sign informed consent.

Exclusion Criteria:

* Pregnant females.
* Mandibular premolars with periodontal pockets greater than 5 mm or greater than grade I mobility.
* Patients have a positive history of antibiotic use or analgesic use within the past week or required antibiotic premedication for dental treatment (such as prosthetic joint prophylaxis).
* Patients have teeth that have been previously accessed.
* Teeth with extensive crown destruction by caries that will not permit rubber dam placement.
* Teeth associated with acute periapical abscess, swelling or a fistulous tract.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | up to 72 hours after endodontic treatment
  Postendodontic pain will be measured using Numerical Rating Scale. The Numerical Rating Scale consists of a 0-10 scale, with (0) meaning "no pain" and (10) meaning "the worst pain imaginable". No or mild pain response will be considered success.

SECONDARY OUTCOMES:
Intra-canal bacterial reduction | Bacterial samples will be taken Immediately after root canal instrumentation.
  Intra-canal bacterial count will be measured using a culture technique. The resultant growth will be visually quantified by counting the number of colony forming units per millilitre (CFUs/ mL)

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen Ibrahim, Master's, Principal Investigator — Misr University for Science and Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fatima S, Kumar A, Andrabi SMUN, Mishra SK, Tewari RK. Effect of Apical Third Enlargement to Different Preparation Sizes and Tapers on Postoperative Pain and Outcome of Primary Endodontic Treatment: A Prospective Randomized Clinical Trial. J Endod. 2021 Sep;47(9):1345-1351. doi: 10.1016/j.joen.2021.05.010. Epub 2021 May 29. PMID 34058250
- [Background] Rodrigues RCV, Zandi H, Kristoffersen AK, Enersen M, Mdala I, Orstavik D, Rocas IN, Siqueira JF Jr. Influence of the Apical Preparation Size and the Irrigant Type on Bacterial Reduction in Root Canal-treated Teeth with Apical Periodontitis. J Endod. 2017 Jul;43(7):1058-1063. doi: 10.1016/j.joen.2017.02.004. Epub 2017 May 5. PMID 28483164